CLINICAL TRIAL: NCT03390465
Title: An Open-label, Randomized, Single Dose, 6-Sequence, 3-Period, Cross-over Study to Evaluate a Drug Interaction Between Fixed-dose Combination of Fimasartan/Amlodipine and Hydrochlorothiazide in Healthy Male Subjects
Brief Title: Drug Interaction Study of Fimasartan/Amlodipine/Hydrochlorothiazide in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR1010
Record Dates: First submitted 2017-12-29; First posted 2018-01-04 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Drug-Drug Interaction
MeSH Terms: interventions — fimasartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm1(N=6) (Other): Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
  Interventions: Drug: Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
- Arm2(N=6) (Other): Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
  Interventions: Drug: Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
- Arm3(N=6) (Other): Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
  Interventions: Drug: Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
- Arm4(N=6) (Other): Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
  Interventions: Drug: Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
- Arm5(N=6) (Other): Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
  Interventions: Drug: Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
- Arm6(N=6) (Other): Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
  Interventions: Drug: Fimasartan/Amlodipine combination drug, Hydrochlorothiazide

INTERVENTIONS:
Drug: Fimasartan/Amlodipine combination drug, Hydrochlorothiazide — Fimasartan/Amlodipine combination drug, Hydrochlorothiazide
  Other Names: FAH

SUMMARY:
The purpose of this study is to evaluate the Drug interaction and safety of Fimasartan/Amlodipine and Hydrochlorothiazide in Healthy Male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* A healthy Male adults aged 19-50 years

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease.
* Hypersensitivity to ingredient of IP and other medication, food.
* Participation in any other study within 3months.
* History of whole blood donation within 2months and Apheresis 1month.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Cmax | 0~48hours after medication
  Maximum Concentration of Fimasartan, Amlodipine, Hydrochlorothiazide in plasma

SECONDARY OUTCOMES:
AUCt | 0~48hours after medication
  AUCt(Area under the curve from the dosing time to the last measurable concentration) of Fimasartan, Amlodipine, Hydrochlorothiazide

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Young Kim, Principal Investigator — Inje University
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea